CLINICAL TRIAL: NCT03574415
Title: A Single-center, Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of DWP14012 in Healthy Japanese, Caucasian and Korean
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DWP14012 After Oral Administration in Healthy Japanese, Caucasian and Korean
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DW_DWP14012004
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Japanese_DWP14012 Amg (Experimental): DWP14012 Amg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Japanese_DWP14012 Bmg (Experimental): DWP14012 Bmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Japanese_DWP14012 Cmg (Experimental): DWP14012 Cmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Caucasian_DWP14012 Bmg (Experimental): DWP14012 Bmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Caucasian_DWP14012 Cmg (Experimental): DWP14012 Cmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Korean_DWP14012 Bmg (Experimental): DWP14012 Bmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Korean_DWP14012 Cmg (Experimental): DWP14012 Cmg, tablets, orally, single and multiple administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Placebo (Placebo Comparator): DWP14012 placebo-matching tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP14012 — DWP14012 tablets
  Arms: Caucasian_DWP14012 Bmg; Caucasian_DWP14012 Cmg; Japanese_DWP14012 Amg; Japanese_DWP14012 Bmg; Japanese_DWP14012 Cmg; Korean_DWP14012 Bmg; Korean_DWP14012 Cmg
Drug: Placebo — DWP14012 placebo-matching tablets

SUMMARY:
To evaluate the safety and tolerability of single and multiple ascending oral doses of DWP14012 in healthy Japanese, Caucasian and Korean subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult Caucasian or Japanese or Korean aged 19 to 50 (inclusive) years, at the time of screening.
* Subjects weighing between 50 kg and 90 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit.

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those who have gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* Those who have been Helicobacter pylori positive
* Those whose plasma AST (SGOT) and ALT (SGPT) exceed 1.5 times to the upper limit of the normal range in screening including additional examinations prior to randomization
* Those who have anatomical disability in insertion and maintenance of pH meter catheter

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Cmax | 1d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 5d~10d pre-dose, 11d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96h
  Maximum concentration of DWP14012
Cmax,ss / Cmin,ss | 1d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 5d~10d pre-dose, 11d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96h
  Maximum / Minimum concentration of DWP14012 at steady state
Tmax | 1d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 5d~10d pre-dose, 11d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96h
  Time of maximum concentration
AUClast / AUCinf | 1d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 5d~10d pre-dose, 11d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96h
  Area under the plasma concentration-time curve
T1/2 | 1d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 5d~10d pre-dose, 11d pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96h
  Elimination half-life
Percentage of total time that the intragastric pH was above 4 | Day 1
  After single administration of the investigational products, 24hr gastric pH monitoring started.
Percentage of total time that the intragastric pH was above 4 | Day 7
  After single administration of the investigational products, 24hr gastric pH monitoring started.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea